CLINICAL TRIAL: NCT00713518
Title: Phase II Open Label Multicenter, Prospective, Randomized, Age Related Macular Degeneration, Comparator Controlled Study Evaluating PF-04523655 Versus Ranibizumab In The Treatment Of Subjects With Choroidal Neovascularization (MONET Study).
Brief Title: Phase II Open Label Multicenter Study For Age Related Macular Degeneration Comparing PF-04523655 Versus Lucentis In The Treatment Of Subjects With CNV (MONET Study).
Acronym: MONET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quark Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B0451001
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD Age Related Macular Degeneration Choroidal Neovascularization Monet
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; PF-04523655

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 ranibizumab (Active Comparator): 0.5 mg ranibizumab intravitreal injection given every 4 weeks from baseline to Week 12
  Interventions: Drug: 0.5 mg ranibizumab
- Arm 2 ranibizumab and PF-04523655 (Experimental): 0.5 mg ranibizumab given by intravitreal injection at baseline followed by 3 mg PF-04523655 given by intravitreal injection every 2 weeks from Week 4 to Week 12
  Interventions: Drug: 0.5 mg ranibizumab; Drug: 3 mg PF-04523655
- Arm 3 ranibizumab and PF-04523655 (Experimental): 0.5 mg ranibizumab given by intravitreal injection at baseline followed by 1 mg PF-04523655 given by intravitreal injection evey 4 weeks to Week 12
  Interventions: Drug: 0.5 mg ranibizumab; Drug: 1 mg PF-04523655
- Arm 4 ranibizumab and PF-04523655 (Experimental): 0.5 mg ranibizumab given by intravitreal injection at baseline followed by 3 mg of PF-04523655 given by intravitreal injection every 4 weeks from Week 4 to Week 12
  Interventions: Drug: 0.5 mg ranibizumab; Drug: 3 mg PF-04523655
- Arm 5 ranibizumab and PF-04523655 (Experimental): 0.5 mg ranibizumab given by intravitreal injection at baseline followed by 1 mg of PF-04523655 (30 minutes later) given in combination every 4 weeks from baseline to Week 12
  Interventions: Drug: 0.5 mg ranibizumab; Drug: 1 mg PF-04523655

INTERVENTIONS:
Drug: 0.5 mg ranibizumab
  Other Names: Lucentis
Drug: 3 mg PF-04523655
  Arms: Arm 2 ranibizumab and PF-04523655; Arm 4 ranibizumab and PF-04523655
Drug: 1 mg PF-04523655
  Arms: Arm 3 ranibizumab and PF-04523655; Arm 5 ranibizumab and PF-04523655

SUMMARY:
The aim of the study is to evaluate whether PF-04523655 is effective in the treatment of neovascular/wet AMD and at which dose.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 50 years or older with active primary or recurrent subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD). Active CNV is defined as any leakage detected on FFA or OCT. Note: Female subjects 50- 60 years of age must be amenorrheic for at least 2 years and have a serum FSH level within the laboratory reference range for postmenopausal women
* The total area of CNV (including both classic and occult components) encompassed within the lesion must be 50% or more of the total lesion area.
* The total lesion size ≤12 disc areas.
* Best corrected visual acuity using ETDRS protocol of 20/40 to 20/320 (letter score ≤73) in the study eye at the screening visit.
* Best corrected visual acuity score in the fellow eye of 20/400 or better (letter score of ≥19) at the Screening Visit. Note: Only one eye will be treated (study eye) through the duration of the study. In the event both eyes are eligible for study entry the study eye should be selected by the investigator and subject. The non-study eye may be treated with an approved AMD therapy
* Subject has retinal central subfield thickness ≥250µm measured using Stratus OCT.

Exclusion Criteria:

* Prior treatment with verteporfin photodynamic therapy, external-beam radiation therapy, or transpupillary thermotherapy in the study eye
* Previous subfoveal focal laser photocoagulation in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1 month preceding Baseline
* History of vitrectomy, submacular surgery or other surgical intervention for AMD in the study eye
* Previous participation in any studies with investigational drugs or treatments administered 1 month preceding Baseline visit such as systemic glucocorticoids, ocular or periocular steroids (eg, triamcinolone, anecortave acetate), anti-angiogenic drugs such as pegaptanib (Macugen), ranibizumab (Lucentis), bevacizumab (Avastin) in the study eye
* Subretinal hemorrhage in the study eye that involves the fovea, if the size of the hemorrhage is either 50% or more of the total lesion area or 1 or more disc areas in size
* CNV in either eye of other etiology, eg, ocular histoplasmosis, trauma, or pathologic myopia
* Presence of subfoveal scarring
* Retinal pigment epithelial tear involving the macula in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Mean change in the best corrected visual acuity score measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol by Week 16 | Week 16

SECONDARY OUTCOMES:
Percent of subjects gaining >/=15 letters in the best corrected visual acuity score at 16 weeks compared to Baseline, as measured using the ETDRS protocol | Week 16
Mean change from Baseline over time (16 weeks) in the best corrected visual acuity score, as measured using the ETDRS protocol | Week 16
Incidence and severity of ocular adverse events identified by ophthalmic examination and or spontaneously reported | Week 48
Change from Baseline to Weeks 4,8, 12, and 16 in retinal central subfield thickness and retinal lesion thickness assessed by OCT | Week 16
Incidence and severity of systemic adverse events identified by physical examination, changes in vital signs, clinical laboratory abnormalities and or spontaneously reported | Week 48
Change from Baseline in lesion size on FFA at Week 16 | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (7):
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Winter Haven, Florida
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Austin, Texas
- Austria (2):
  - Pfizer Investigational Site, Linz
  - Pfizer Investigational Site, Vienna
- Pfizer Investigational Site, Glostrup Municipality, Denmark
- Pfizer Investigational Site, Hong Kong, Hong Kong
- India (4):
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Navrangpura, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Coimbatore, Tamil Nadu
  - Pfizer Investigational Site, New Delhi
- Israel (5):
  - Pfizer Investigational Site, Kfar Saba
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel Aviv
  - Pfizer Investigational Site, Tel Litwinsky
  - Pfizer Investigational Site, Ẕerifin
- Philippines (3):
  - Pfizer Investigational Site, Makati City
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Quezon City
- Pfizer Investigational Site, Seoul, South Korea
- Spain (3):
  - Pfizer Investigational Site, Alicante, Alicante
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Valencia, Valencia
- Pfizer Investigational Site, Taipei, Taiwan
- Pfizer Investigational Site, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0451001&StudyName=Phase%20II%20Open%20Label%20Multicenter%20Study%20For%20Age%20Related%20Macular%20Degeneration%20Comparing%20An%20Investigational%20Drug%20PF-04523655%20Versus%20Lucentis%20I